CLINICAL TRIAL: NCT00939094
Title: A Phase IIa, Double-Blind, Randomised, Parallel-Group, Multi-Centre Study to Evaluate the Analgesic Efficacy of 28 Days Oral Administration of AZD2066 Compared to Placebo in Peripheral Neuropathic Pain Patients With Mechanical Hypersensitivity
Brief Title: AZD2066 Neuropathic Pain - Mechanical Hypersensitivity
Acronym: NP-MH
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D0475C00016
Record Dates: First submitted 2009-07-13; First posted 2009-07-14 (Estimated); Results first posted 2012-09-27 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2012-08

CONDITIONS: Neuropathic Pain; Mechanical Hypersensitivity
Keywords: Pain, Mechanical Hypersensitivity; Allodynia; Efficacy; analgesia; Neuropathic
MeSH Terms: conditions — Neuralgia; Pain; Hyperalgesia; Agnosia | interventions — AZD2066

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- A (Experimental)
  Interventions: Drug: AZD2066
- B (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD2066 — Capsule, once daily
  Arms: A
Drug: Placebo — Capsule, once daily
  Arms: B

SUMMARY:
The purpose of this study is to investigate if 28 days of treatment with AZD2066 compared to placebo can relieve the pain arising from the nervous system when the patients are touched by something that should not cause pain or have severe pain when they are touched by something that should only cause a little pain.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures.
* Male or non-fertile females
* Painful symptoms due to neuropathic pain for a period of 3 months to 5 years, associated with mechanical allodynia and/or punctate hyperalgesia.

Exclusion Criteria:

* Other pain that may confound assessment of neuropathic pain.
* Diagnosis of any severe neurological disease.
* History of significant psychiatric disease/condition and/or history of psychotic disorders among first degree relatives.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2009-08; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Biljana Lilja, Study Director — AstraZeneca R&D Södertälje151 85 Södertälje, Sweden; Brett Stacey, Principal Investigator — Oregon Health and Science University Comprehensive Pain Clinic, Portland, OR 97239, USA
Locations (38):
- United States (38):
  - Research Site, Tucson, Arizona
  - Research Site, Los Angeles, California
  - Research Site, Sacramento, California
  - Research Site, San Francisco, California
  - Research Site, Walnut Creek, California
  - Research Site, Boulder, Colorado
  - Research Site, Atlantis, Florida
  - Research Site, Aventura, Florida
  - Research Site, Clearwater, Florida
  - Research Site, Fort Myers, Florida
  - Research Site, Orlando, Florida
  - Research Site, Palm Beach Gardens, Florida
  - Research Site, Sarasota, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Sunrise, Florida
  - Research Site, Canton, Georgia
  - Research Site, Marietta, Georgia
  - Research Site, Evansville, Indiana
  - Research Site, New Orleans, Louisiana
  - Research Site, Brockton, Massachusetts
  - Research Site, Bingham Farms, Michigan
  - Research Site, Las Vegas, Nevada
  - Research Site, Reno, Nevada
  - Research Site, Lumberton, New Jersey
  - Research Site, Willingboro, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Jacksonville, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Kettering, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Bridgeville, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Irving, Texas
  - Research Site, Lexington, Texas
  - Research Site, Longview, Texas
  - Research Site, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter study was conducted between August 2009 and November 2010 in the United States.
Pre-assignment Details: The study had an enrolment phase of up to 35 days (including washout and baseline periods), a 28-day treatment phase, and a follow-up phase of 7 days (for men and women not of childbearing potential) or 28 days (for women of childbearing potential). Patients randomized to AZD2066 received AZD2066 12 mg from Days 1 to 4 and 18 mg from Days 5 to 28.
Groups:
- A - AZD2066: AZD2066, 12 mg capsule
- 2 - Placebo: Placebo, capsule
Period: Overall Study
Arm/Group | A - AZD2066 | 2 - Placebo
Started | 42 | 45
Completed | 28 | 35
Not Completed | 14 | 10
Not completed — Adverse Event | 9 | 0
Not completed — Withdrawal by Subject | 1 | 6
Not completed — Lost to Follow-up | 1 | 1
Not completed — Eligibility criteria not fulfilled | 2 | 0
Not completed — Severe non-compliance to protocol | 0 | 1
Not completed — Study stopped by sponsor | 0 | 2
Not completed — Abnormal ECG findings | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A - AZD2066 | 2 - Placebo | Total
Number analyzed (Participants) | 42 | 45 | 87
Age Continuous [Mean (Standard Deviation); unit: years] | 58.1 (9.25) | 59.3 (14.31) | 58.7 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 18 | 42
  Male | 18 | 27 | 45

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Numerical Rating Scale (NRS) Pain Score From Baseline to Last 5 Days on Treatment
Description: Mean pain intensity for 5-day baseline period (morning Day -5 to evening Day-1) and mean pain intensity for last 5 days on treatment (ie, last dose day and the 4 preceding calendar days) was calculated based on the NRS scale (0-10). 0=No pain, 10=Worst pain imaginable.
Time Frame: Change in mean pain intensity from 5-day baseline to the last 5 days on treatment, measure twice daily with NRS (12-hour recall)
Measure: Least Squares Mean (Standard Error); unit: Scores (units) on NRS
Arm/Group | A - AZD2066 | 2 - Placebo
Number analyzed (Participants) | 30 | 38
Scores (units) on NRS | -2.14 (0.358) | -1.26 (0.337)

2. Secondary Outcome: Patients With ≥30% Reduction From Baseline in NRS Pain Intensity Score (Responder Rate) at Day 28
Description: NRS pain intensity score reduction=(change from baseline at Day 28/baseline)*100 Responder=pain intensity score reduction ≥30% (yes/no)? Responder rate=(no. of responders/total no. of patients)*100
Time Frame: 28 days
Measure: Number; unit: Participants
Arm/Group | A - AZD2066 | 2 - Placebo
Number analyzed (Participants) | 30 | 38
Participants | 16 | 10

3. Secondary Outcome: Patients With ≥50% Reduction From Baseline in NRS Pain Intensity Score (Responder Rate) at Day 28
Description: Pain intensity score reduction=(change from baseline Day 28/baseline)*100 Responder=pain intensity score reduction ≥50% (Yes/No)? Responder rate=(no. of responders/total no. of patients)*100
Time Frame: 28 days
Measure: Number; unit: Participants
Arm/Group | A - AZD2066 | 2 - Placebo
Number analyzed (Participants) | 30 | 38
Participants | 10 | 5

4. Secondary Outcome: Patients With Patient Global Impression of Change (PGIC) Score of at Least "Much Improved" (Responder Rate) at Day 28
Description: PGIC scale ranges from 1-7 where 1=Very much improved and 7=Very much worse Responder=Patient with a response of " much improved" or "very much improved" Responder rate=(no. of responders/total no. of patients)*100
Time Frame: 28 days
Measure: Number; unit: Patients
Arm/Group | A - AZD2066 | 2 - Placebo
Number analyzed (Participants) | 30 | 38
Patients | 10 | 10

5. Secondary Outcome: Change in Short Form McGill Pain Questionnaire (SF-MPQ) Sensory Index From Baseline to Day 28
Description: Sensory index=sum of the intensity scale values of the words chosen for the descriptors 1-11 in the questionnaire. Range of scores for the sensory index=0-33 (higher score represents a worse condition).
  Change from baseline (measured prior to randomization) to Day 28 was calculated.
Time Frame: 28 days
Measure: Least Squares Mean (Standard Error); unit: Scores (units) on SF-MPQ Sensory Index
Arm/Group | A - AZD2066 | 2 - Placebo
Number analyzed (Participants) | 30 | 38
Scores (units) on SF-MPQ Sensory Index | -6.39 (1.278) | -3.98 (1.188)

6. Secondary Outcome: Change in SF-MPQ Affective Index From Baseline to Day 28
Description: Affective index=sum of the intensity scale values of the words chosen for the descriptors 12-15 in the questionnaire. Range of scores for the affective index=0-12 (higher score represents a worse condition).
  Change from baseline (measured prior to randomization) to Day 28 was calculated.
Time Frame: 28 days
Measure: Least Squares Mean (Standard Deviation); unit: Scores (units) on SF-MPQ Affective Index
Arm/Group | A - AZD2066 | 2 - Placebo
Number analyzed (Participants) | 30 | 38
Scores (units) on SF-MPQ Affective Index | -1.1 (0.52) | -0.9 (0.50)

7. Secondary Outcome: Change in Brief Pain Inventory-Short Form (BPI-SF) Pain Severity From Baseline to Day 28
Description: Change from baseline (measured prior to randomization) to Day 28 was calculated for the pain severity (mean of 4 intensity items). Each intensity item is recorded on a NRS 0-10, where 0=No Pain and 10=Pain as bad as you can imagine.
Time Frame: 28 days
Measure: Least Squares Mean (Standard Error); unit: Scores (units) on BPI-SF pain severity
Arm/Group | A - AZD2066 | 2 - Placebo
Number analyzed (Participants) | 30 | 38
Scores (units) on BPI-SF pain severity | -2.12 (0.385) | -1.25 (0.360)

8. Secondary Outcome: Change in BPI-SF Pain Interference From Baseline to Day 28
Description: Change from baseline (measured prior to randomization) to Day 28 was calculated for pain interference (mean of 7 interference items). Each interference item is recorded on a NRS 0-10, where 0=No interference and 10=Interferes completely.
Time Frame: 28 days
Measure: Least Squares Mean (Standard Error); unit: Scores on BPI-SF pain interference
Arm/Group | A - AZD2066 | 2 - Placebo
Number analyzed (Participants) | 30 | 38
Scores on BPI-SF pain interference | -1.98 (0.376) | -1.72 (0.360)

ADVERSE EVENTS:
Arm/Group | A - AZD2066 | 2 - Placebo
Serious Adverse Events (participants affected / at risk) | 1/42 | 0/44
Other Adverse Events (participants affected / at risk) | 30/42 | 15/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A - AZD2066 (N=42) | 2 - Placebo (N=44)
Psychotic Disorder (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | A - AZD2066 (N=42) | 2 - Placebo (N=44)
Dizziness (Nervous system disorders) | 10 | 3
Headache (Nervous system disorders) | 7 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 2
Diarrhea (Gastrointestinal disorders) | 3 | 2
Insomnia (Psychiatric disorders) | 3 | 1
Paraesthesia (Nervous system disorders) | 3 | 0
Somnolence (Nervous system disorders) | 3 | 0
Constipation (Gastrointestinal disorders) | 0 | 3

LIMITATIONS AND CAVEATS:
Early termination of study for safety reasons leading to fewer subjects analyzed than originally planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication or presentation with respect to the study until the earlier of 1) publication of the first Multi-Center Publication and 2) the second anniversary of the completion, or termination of the study.

Sponsor to review at least 60 days prior submission. Sponsor can withhold material for submission for additional 90 days